CLINICAL TRIAL: NCT03867448
Title: The Evaluation and Management of Endocrine-Related Conditions and Physiology
Brief Title: Study of Endocrine-Related Conditions and Physiology
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190066; 19-DK-0066
Record Dates: First submitted 2019-03-07; First posted 2019-03-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-27

CONDITIONS: Endocrine Disease
Keywords: Adrenal Gland; Pituitary; Natural History
MeSH Terms: conditions — Endocrine System Diseases; Pituitary Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with Endocrine Disorder: Adults referred to NIH with possible endocrine conditions

SUMMARY:
Background:

Endocrine disorders involve changes to glands that produce hormones. Hormones are released by these glands into the blood so they can direct the function of other tissues in the body. Researchers want to study people who may have endocrine disorders. They want to learn more about the conditions that affect endocrine glands.

Objective:

To study adults with a variety of endocrine disorders for research and physician education.

Eligibility:

Adults ages 18 and older who have an endocrine or metabolic-related disorder

Healthy volunteers 18 and older

Design:

Participants will be screened with a review of their medical records.

Participants will have a physical exam and medical history.

The length of the study and the schedule will vary by participant. Tests may include:

Blood and urine tests

Stool and saliva samples

Imaging studies: Participants will lie on a table while a machine takes pictures of the body. They may be injected with a substance to make their organs more visible in the pictures.

Tests of endocrine tissue function

Consultation with other specialists

Sleep study

Medical photographs

Participants may be treated for their endocrine disorder. This could include:

Surgery. If tissue is removed during surgery, it may be studied.

Radiation

Medicine

Participants may have genetic testing. This will be done with a small amount of blood, cells from a cheek swab, or saliva.

Sponsoring Institution: National Institute of Digestive, Diabetes and Kidney Disease

DETAILED DESCRIPTION:
Study Description:

This study allows the NIH Intramural Endocrinology Training Program (IETP) to follow or provide evaluation, treatment and or interventions to certain eligible subjects.

Objectives:

1. To provide a repository of data and samples obtained during the course of clinical care to allow for future research.
2. To add value to the IEFP training program by maintaining a diverse group of endocrine conditions seen at the NIH.
3. To provide a vehicle by which pilot studies of endocrine physiology can be initiated.
4. To identify prismatic cases that deviate from known presentations or responses to treatment.
5. To evaluate the safety and results from adrenal venous sampling using a modified catheter with side hole placement.

Endpoints:

1. Data from standard of care evaluation and management.
2. Adverse events during and after adrenal vein sampling; cortisol and aldosterone results from the sampling.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all the following criteria:

* Adult men and women age 18 years or older.
* Known or suspected endocrine disorders requiring clinical screening, management and/or treatment and follow-up.
* Stated willingness to comply with all study procedures and availability for the duration of the study

EXCLUSION CRITERIA:

* Unstable participants and participants with severe organ failure, or those with a condition or medical treatment that may affect/limit the endocrine work-up and exhaust Clinical Center, IETP resources will be excluded if appropriate.
* Inability of a subject to adhere to a proposed schedule of visits.
* Inability to provide informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any adult with a potential endocrine disorder; the types of disorders may vary to ensure that there is an adequate case mix of diagnoses for the training program.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-03-27 (Actual); Primary Completion 2036-01-01 (Estimated); Study Completion 2036-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis/Treatment | variable
  determination of diagnosis and/or treatment of an endocrine disorder

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
WE currently have no plan to share this data, but in the future may consider sharing of this data for analysis with collaborators of with other expertise.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-DK-0066.html